CLINICAL TRIAL: NCT04660695
Title: Serie de Casos Prospectiva de Gastroenteroanastomosis Guiada Por Ecoendoscopia Para la obstrucción al Vaciado gástrico en Neoplasias Avanzadas Mediante la técnica Del Drenaje Nasobiliar
Brief Title: Nasobiliary Drain Assisted EUS-guided Gastroenterostomies in Unresectable Malignant Gastric Outlet Obstruction
Acronym: PENGUIN
Status: Completed | Type: Observational
Sponsor: Hospital del Rio Hortega (Other)
Collaborators: Hospital General Universitario de Alicante (Other); Clinica Universidad de Navarra, Universidad de Navarra (Other); Complejo Hospitalario de Navarra (Other); Christian Medical College, Vellore, India (Other)
Responsible Party: Principal Investigator, Francisco Javier Garcia Alonso, Md PhD, Hospital del Rio Hortega
Other Study IDs: PI152-19
Record Dates: First submitted 2020-11-23; First posted 2020-12-09 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Gastric Outlet Obstruction; Gastric Cancer; Pancreatic Cancer
MeSH Terms: conditions — Gastric Outlet Obstruction; Stomach Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Group 1: Patients included will undergo an EUS-guided gastroenterostomy with a 15x10mm or a 20x10mm lumen apposing metal Stent (Axios, Boston Scientific, Mass).
  Interventions: Device: EUS-guided gastroenterostomy

INTERVENTIONS:
Device: EUS-guided gastroenterostomy — Firstly, un upper digestive endoscopy is performed with a conventional gastroscope. A guidewire is passed through the malignant lesion causing the gastric outlet obstruction. Once the guidewire is located in the distal duodenum/proximal jejunum, a nasobiliary drain (Nasal Biliary Drainage Sets, Cook medical, Indiana) is advanced over the guidewire until its distal end is placed in the distal duodenum/jejunum. At this point the gastroscope is substituted by a therapeutic echoendoscope. With the echoendoscope in place, the target bowel loop is filled with saline combined with methilene blue and radiopaque contrast. The echoendoscope is used to identify the target bowel loop. AFter identifying the target, a lumen apposing metal stent (Axios, Boston Scientific, Massachusetts) is deployed across the gastric and bowel using its electrocautery enhanced deployment device.
  Other Names: AXIOS™ Stent and Electrocautery Enhanced Delivery System (Boston Scientific, Mass)

SUMMARY:
Gastric outlet obstruction in malignant disease appears when the tumor affects the gastroduodenal area, precluding the passage of food into the small bowel. This condition severely affects the quality of life. In patients with unresectable tumors, there are various available treatments:a surgical bypass connecting the stomach to the small bowel, placing a stent through the tumor to widen the passage and creating a gastrointestinal bypass with a lumen apposing metal stent. These stents are deployed with an echoendoscope, which allows to identify a small bowel loop and to deploy the stent, connecting the small bowel and the stomach. This is called a EUS-guided gastroenterostomy (EUS-GE).

EUS-GE is a rather novel procedure. Various techniques to create EUS-GE have been proposed. In this study, the investigators will retrieve data from the procedure and during the thirty following days from consecutive patients undergoing an EUS-GE. The objectives of the study are:

* To perform a detailed step by step description of the nasobiliary drain assisted EUS-GE
* To describe the adverse events encountered
* To describe the proportion of clinical and technical success
* To assess its impact on the patients' quality of life.
* To assess the evolution of the oral intake during the first month after the procedure

DETAILED DESCRIPTION:
DESIGN

Prospective multicenter case series

AIMS

Primary aim To describe the proportions of technical and clinical success. To describe different variants in the nasobiliary drain assissted EUS-GE technique, offering a detailed step by step description of the procedure performance by different endoscopists

Secondary aims:

To describe the adverse encountered, their severity according to ASGE standards and their management.

To describe the time elapsed between the procedure and the initial oral intake.

To describe the evolution of the oral intake during the first month after the procedure To assess the impact of the operators experience on procedure times, adverse events and technical issues.

To assess the impact of the procedure on the quality of life of the participating patients.

STUDY POPULATION

All consecutive patients over 18 years of age receiving a nasobiliary drain assisted EUS-GE for unresectable malignant GOO are eligible to participate in this study. Patients with a previous gastroduodenal surgery, a previous endoscopic or surgical treatment for GOO, a simultaneous malignant biliary obstruction requiring endoscopic treatment, a distal bowel obstruction, ascites grade 2 or superior, uncorrectable coagulation disorders (INR>1,5) or severe thrombocytopenia (<50000 platelets/mm3). or unable to understand the questionnaires will be excluded.

INTERVENTION

At inclusion

Informed consent will be obtained. A clinical interview and a physical examination will be performed. TheEuropean Organization for Research and Treatment of Cancer QoL Questionnaire Core 30 (EORTC-QLQ-C30), which includes 30 items covering a global health status scale, five functional scales and ten symptom scales will be assessed in a telephone interview.

Endoscopic procedure

All procedures will be performed under sedation. An assistant endoscopist or research nurse will retrieve all data regarding the procedure. Firstly, un upper digestive endoscopy is performed with a conventional gastroscope. A guidewire is passed through the malignant lesion causing the gastric outlet obstruction. Once the guidewire is located in the distal duodenum/proximal jejunum, a nasobiliary drain (Nasal Biliary Drainage Sets, Cook medical, Indiana) is advanced over the guidewire until its distal end is placed in the distal duodenum/jejunum. At this point the gastroscope is substituted by a therapeutic echoendoscope. With the echoendoscope in place, the target bowel loop is filled with saline combined with methilene blue and radiopaque contrast. The echoendoscope is used to identify the target bowel loop. AFter identifying the target, a lumen apposing metal stent (Axios, Boston Scientific, Massachusetts) is deployed across the gastric and bowel using its electrocautery enhanced deployment device.

Post procedure: Oral liquid intake can be restarted 4h after the procedure in patients presenting no signs or symptoms suggesting any adverse event. Pacients with an adequate tolerance might be discharged.

Follow-up

Clinical telephone interviews by an experienced research nurse will be held via telephone calls 1 day, 7 days and 30 days after the procedure. Oral intake and adverse events will be assessed every visit. Thirty days after the procedure a second evaluation of the EORTC-QLQ-C30 will be performed.

STATISTICAL ANALYSIS

Categorical variables were reported as percentages. Normally distributed continuous variables were reported as the mean with the standard deviation values. Non-normally distributed continuous variables were reported as the median and interquartile range. The EORTC QLQ-C30 descriptive analysis was performed with a specifically programmed Stata command (10). Variables regarding the procedure step by step analysis will only undergo a descriptive analysis. Differences between the different outcomes of the EORTC-QLQ-C30 will be assessed using linear mixed models with fixed effects for baseline values, and interaction with oncological treatment. The statistical analysis will be performed using the Stata package (StataCorp. 2013, College Station, Texas).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* unresectable malignant gastric outlet obstruction
* Undergoing placement of nasobiliary drain assisted EUS-GE

Exclusion Criteria:

* Previous gastroduodenal surgery
* Previous endoscopic or surgical treatment for gastric outlet obstruction
* Simultaneous biliary obstruction (malignant or benign) requiring endoscopic treatment
* Simultaneous upper digestive tract disease requiring endoscopic treatment in the same procedure
* Unable to understand the questionnaires
* Distal bowel obstruction
* Ascites grade 2 or superior
* Uncorrectable coagulation disorders (INR>1,5) or severe thrombocytopenia (<50000 platelets/mm3).
* Active, symptomatic SARS-CoV-2 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients over 18 years of age submitted to any of the participanting center's endoscopy units to receive a nasobiliary drain assisted EUS-GE for unresectable malignant GOO are eligible to participate in this study.
  Patients with a previous gastroduodenal surgery, a previous endoscopic or surgical treatment for GOO, a simultaneous malignant biliary obstruction or unable to understand the questionnaires will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
Technical Success | Day +1
  An adequate stent placement across the GI walls, with one flange in the gastric cavity and the other in the small bowel lumen. It has to be confirmed either fluoroscopically or endoscopically.
Early Clinical Success | Day +7
  Defined as a GOOSS >=2.
Clinical Success | Day +30
  Defined as a GOOSS >=2.

SECONDARY OUTCOMES:
Baseline Gastric outlet obstruction score system (GOOSS) | Baseline
  The GOOSS is a previously defined classification of Gastric outlet obstruction which incudes 4 categories (0-Nil Per Os; 1 liquids only; 2 soft diet; 3 low residue or full diet)
Early Gastric outlet obstruction score system (GOOSS) | day +7
  The GOOSS is a previously defined classification of Gastric outlet obstruction which incudes 4 categories (0-Nil Per Os; 1 liquids only; 2 soft diet; 3 low residue or full diet)
Final Gastric outlet obstruction score system (GOOSS) | day +30
  The GOOSS is a previously defined classification of Gastric outlet obstruction which incudes 4 categories (0-Nil Per Os; 1 liquids only; 2 soft diet; 3 low residue or full diet)
Baseline European Organisation for Research and Treatment of Cancer QoL Questionnaire Core 30 (EORTC-QLQ-C30) | Baseline
  The EORTC-QLQ-C30 is a validated questionnaire (with validated translations in Spanish), which includes 30 items covering a global health status scale, five functional scales and ten symptom scales
Final European Organisation for Research and Treatment of Cancer QoL Questionnaire Core 30 (EORTC-QLQ-C30) | Baseline, day+30
  The EORTC-QLQ-C30 is a validated questionnaire (with validated translations in Spanish), which includes 30 items covering a global health status scale, five functional scales and ten symptom scales
Number of Participants With intraprocedure Treatment-Related Adverse Events as Assessed by the ASGE classification | day+1,
  The ASGE classification is a tool developed to describe and assess the severity of endoscopy related adverse events.
Number of Participants With Early Treatment-Related Adverse Events as Assessed by the ASGE classification | day+7
  The ASGE classification is a tool developed to describe and assess the severity of endoscopy related adverse events.
Number of Participants With Delayed Treatment-Related Adverse Events as Assessed by the ASGE classification | day+30
  The ASGE classification is a tool developed to describe and assess the severity of endoscopy related adverse events.
Recurrent GOO | Day +30
  In patients achieving clinical success in day +7, recurrent GOO is defined as the development of nausea and vomiting and/or a GOOSS<2.
Target bowel loop diameter (mm) | Procedure
  Diameter measured with the EUS of the dilated bowel loop. It should be measured just before placing the stent
Total volume infused (ml) | Procedure
  Volume of saline, methilene blue solution or radiopaque contrast solution instiled to dilate the target bowel loop
Number of patients undergoing balloon dilation | Procedure
  After deploying the stent, it might be dilated with a controlled radial expansion balloon dilator
Type of fluid employed | Procedure
  Three different fluids can be used to dilate the target bowel loop, saline, methilene blue diluted in saline or radiopaque contrast diluted in saline

CONTACTS AND LOCATIONS:
Overall Officials: Carlos de la Serna Higuera, MD, Principal Investigator — Hospital del Rio Hortega
Locations (5):
- Christian Medical College, Vellore, India
- Spain (4):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario Río Hortega, Valladolid

IPD SHARING:
Plan to Share IPD: Undecided
After the study is completed a csv including all study data can be submitted to a repository or made available to applying investigators.

REFERENCES:
- [Derived] Chavarria C, Martin-Alvarez V, Aparicio JR, Subtil JC, Garcia-Alonso FJ, Vila JJ, Martinez-Moreno B, Busto Bea V, de la Serna-Higuera C, Perez-Miranda M. EUS-guided gastroenterostomy using a parallel enteric tube for luminal distension: Prospective multicenter procedural standardization (with video). Endosc Ultrasound. 2025 May-Jun;14(3):129-136. doi: 10.1097/eus.0000000000000123. Epub 2025 Jun 13. PMID 41584027
- [Derived] Garcia-Alonso FJ, Chavarria C, Subtil JC, Aparicio JR, Busto Bea V, Martinez-Moreno B, Vila JJ, Martin-Alvarez V, Sanchez-Delgado L, de la Serna-Higuera C, Perez-Miranda M. Prospective multicenter assessment of the impact of EUS-guided gastroenterostomy on patient quality of life in unresectable malignant gastric outlet obstruction. Gastrointest Endosc. 2023 Jul;98(1):28-35. doi: 10.1016/j.gie.2023.02.015. Epub 2023 Feb 18. PMID 36801458

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-21): https://cdn.clinicaltrials.gov/large-docs/95/NCT04660695/Prot_SAP_000.pdf